CLINICAL TRIAL: NCT05878769
Title: A Phase III Open-Label Extension Study to Evaluate the Long-Term Safety of Astegolimab in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Long-Term Safety of Astegolimab in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB43374
Record Dates: First submitted 2023-05-19; First posted 2023-05-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — astegolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Extension (Experimental): Eligible participants from parent studies GB43311 and GB44332 will receive subcutaneous (SC) astegolimab every 2 weeks (Q2W) until the end of the study
  Interventions: Drug: Astegolimab

INTERVENTIONS:
Drug: Astegolimab — Participants will receive SC astegolimab Q2W

SUMMARY:
The purpose of this study is to assess the long-term safety and to explore the efficacy of astegolimab in participants with chronic obstructive pulmonary disease (COPD) who have completed the 52-week placebo-controlled treatment period in parent studies GB43311 or GB44332.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the 52-week treatment period in either parent GB43311 or GB44332

Exclusion Criteria:

* Withdrawal of consent and/or premature discontinuation from parent study
* Any permanent discontinuation of study drug in parent study
* Significant non-compliance in the parent study, specifically defined as missing scheduled visits, per investigator's judgment
* Any new diagnosis of asthma according to the Global Initiative for Asthma guidelines or other accepted guidelines since enrolling in the parent study
* Any new clinically significant pulmonary disease other than COPD (e.g., pulmonary fibrosis, sarcoidosis, chronic pulmonary embolism or primary pulmonary hypertension, alpha-1-antitrypsin deficiency) since enrolling in the parent study
* Any new unstable cardiac disease, myocardial infarction, or New York Heart Association Class III or IV heart failure since enrolling in the parent study

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of all adverse events (AEs) | Up to 12 weeks after last dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (478):
- United States (68):
  - UAB Lung Health Center, Birmingham, Alabama
  - SEC Clinical Research LLC - Dothan 2 - ClinEdge - PPDS, Dothan, Alabama
  - Jasper Summit Research LLC, Jasper, Alabama
  - Pulmonary Associates of Mobile PC, Mobile, Alabama
  - Pulmonary Associates Deer Valley Office, Phoenix, Arizona
  - AES - DRS - Synexus Clinical Research US, Inc. - Tucson, Tucson, Arizona
  - Kern Allergy and Medical Research, Bakersfield, California
  - Cadena Care Institute, LLC, Poway, California
  - Apex Clinical Research, San Diego, California
  - St Francis Medical Institute ClinEdge PPDS, Clearwater, Florida
  - Finlay Medical Research Corporation, Greenacres City, Florida
  - Flourish Research - Leesburg - PPDS, Leesburg, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - San Marcus Research Clinic Inc., Miami, Florida
  - Finlay Medical Research Corporation, Miami, Florida
  - Oceane7 Medical & Research Center, Inc., Miami, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Diverse Clinical Research, LLC, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Florida Institute for Clinical Research, LLC, Orlando, Florida
  - Flourish Research - Orlando - PPDS, Winter Park, Florida
  - Pivotal Research Solutions, Stonecrest, Georgia
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - ASHA Clinical Research - ClinEdge - PPDS, Hammond, Indiana
  - Best Clinical Trials, New Orleans, Louisiana
  - Paul A. Shapero, MD, PA, Bangor, Maine
  - Exordia Medical Research, Inc., Fall River, Massachusetts
  - Pulmonary Research Institute of Southeast Michigan, Farmington Hills, Michigan
  - Flushing Road Internal Medicine and Pediatrics - F, Flint, Michigan
  - Revive Research Institute, Southfield, Michigan
  - Oakland Medical Research, Troy, Michigan
  - The Lung Research Center, Chesterfield, Missouri
  - Hannibal Regional Healthcare System HRMG Hannibal, Hannibal, Missouri
  - Midwest Chest Consultants, Saint Charles, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Midwest Clinical Research LLC, St Louis, Missouri
  - The Machuca Foundation Inc, Las Vegas, Nevada
  - Sierra Clinical Research - ClinEdge - PPDS, Las Vegas, Nevada
  - Renown Regional Medical Center Hospital, Reno, Nevada
  - AES - DRS - Synexus Clinical Research US, Inc. - New York, New York, New York
  - American Health Research Inc., Charlotte, North Carolina
  - Research Carolina Elite, Denver, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Pulmonix LLC, Greensboro, North Carolina
  - Carolina Research Center, Shelby, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - OK Clinical Research, Edmond, Oklahoma
  - The Oregon Clinic., Portland, Oregon
  - Clinical Research Associates Of Central Pa , Llc, DuBois, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allergy & Clinical Immun Assoc, Pittsburgh, Pennsylvania
  - Medtrial, LLC, Columbia, South Carolina
  - Velocity Clinical Research - Gaffney - PPDS, Gaffney, South Carolina
  - Lowcountry Lung and Critical Care, North Charleston, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Tennessee Comprehensive Lung & Sleep Center, Hendersonville, Tennessee
  - South Texas Medical Research Institute, Inc., dba TTS Research ? ClinEdge ? PPDS, Boerne, Texas
  - Corsicana Medical Research, Corsicana, Texas
  - Trio Clinical Trials, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Pulmonary Medicine Associates, PA - Biopharma Informatic, LLC, Houston, Texas
  - Metroplex Pulmonary and Sleep Medicine Center, McKinney, Texas
  - Sherman Clinical Research - ClinEdge - PPDS, Sherman, Texas
  - Vermont Lung Center at the University of Vermont, Colchester, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Western Washington Medical Group, Everett, Washington
  - Allergy Asthma and Sinus Center-Greenfield, Greenfield, Wisconsin
- Argentina (40):
  - Centro Medico Capital, La Plata, Buenos Aires
  - Consultorios Medicos Organizacion de Buen Ayre SRL, Buenos Aires
  - Centro de Investigaciones Clínicas Belgrano, Buenos Aires
  - Fundacion Cidea, Buenos Aires
  - Fundacion Faicep, Buenos Aires
  - Instituto de Investigaciones En Alergia Y Enfermedades Respiratorias, Buenos Aires
  - AES - AS - Glenny Corp. S.A. Buenos Aires, Buenos Aires
  - CARE - Centro de Alergia y Enfermedades Respiratorias, CABA
  - Nexo Salud Investigacion Clinica - Riobamba 429, Ciudad Autonoma Buenos Aires
  - CINME S.A. ? Centro de Investigaciones Metabolicas - Rx Trials LLC, Ciudad Autonoma Buenos Aires
  - Centro Médico Dra de Salvo, Ciudad Autonoma Buenos Aires
  - Centro de Medicina Respiratoria, Concepción del Uruguay
  - Sanatorio de la Canada, Córdoba
  - Instituto de Medicina Respiratoria, IMeR, Córdoba
  - Centro Privado de Medicina Respiratoria, Entre Ríos
  - Framingham Centro Medico, La Plata
  - Centro Platense en Investigaciones Respiratorias, La Plata
  - Centro de Especialidades Medicas Lobos, Lobos
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Instituto de Investigaciones Clinicas-Mar del Plata, Mar del Plata
  - Instituto Ave Pulmo, Mar del Plata
  - Centro Medico Dharma, Mendoza
  - Fundacion Scherbovsky, Mendoza
  - INSARES, Mendoza, Mendoza City
  - Centro Respiratorio Quilmes, Quilmes
  - Sala de primeros auxilios Alberto Mignaburu, Ranelagh, Berazategui
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
  - Sanatorio Parque de Rosario, Rosario
  - Instituto Medico Fundacion Grupo Colaborativo Rosario Investigacion y Prevencion Medica, Rosario
  - Servicio de Investigacion de Patologias Alergicas-Instituto ABC, Rosario
  - Centro Medico IPAM, Rosario
  - Centro Médico Respire, San Fernando
  - Instituto De Patologias Respiratorias, San Miguel de Tucumán
  - Centro Integral de Medicina Respiratoria (CIMER), San Miguel de Tucumán
  - Centro Modelo de Cardiologia, San Miguel de Tucumán
  - Centro Medico San Nicolas Grupo Orono, San Nicolás de los Arroyos
  - CEPROSS- Centro Profesional San Salvador, San Salvador
  - Instituto Del Buen Aire, Santa Fe
  - Centro de Diagnostico Y Rehabilitacion, Santa Fe
  - Instituto De Enfermedades Respiratorias E Investigacion Medica, Villa Vatteone
- Australia (4):
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Institute for Respiratory Health Inc, Midland, Western Australia
  - TrialsWest Pty Ltd, Spearwood, Western Australia
- Austria (2):
  - Ordination Dr. Robert Voves, Feldbach
  - Ordination fur Lungenkrankheiten, Linz
- Belgium (10):
  - AZ Sint-Jan Brugge-Oostende, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Antwerp University Hospital, Edegem
  - Private Practice Dr Jean Benoit Martinot, Erpent
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - AZ Sint-Maarten, Mechelen
  - AZ Delta, Roeselare
  - Office of Marc De Meulemeester, Thuin
  - CHU UCl Namur asbl - Site Godinne, Yvoir
- Brazil (5):
  - LMK Servicos Medicos SS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo, São Paulo
  - IBPCLIN Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
- Bulgaria (25):
  - MHAT Knyaginya Klementina Sofia EAD, Sofia, Sofia-Grad
  - Diagnostic-Consultative Center Aleksandrovska EOOD, Sofia, Sofia-Grad
  - Multiprofile Hospital for Active Treatment Puls AD PPDS, Blagoevgrad
  - Multiprofile Hospital For Active Treatment Sveta Ekaterina - Dimitrovgrad EOOD, Dimitrovgrad
  - Medical Centre "Asklepii", OOD, Dupnitsa
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases - Haskovo EOOD, Haskovo
  - Medical Centre Pratia EOOD branch Lovech, Lovech
  - Medical Center Hera EOOD, Montana
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases-Dr.Nikola Penchev-Paza, Pazardzhik
  - Specialized Hospital for Active Treatment of Pulmonary Diseases- Pernik EOOD, Pernik
  - Medical center Medconsult Pleven OOD, Pleven
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Medical center Unimed EOOD, Plovdiv
  - Multiprofile Hospital for Active Treatment Shumen, Shumen
  - Multiprofile Hospital for Active Treatment - Silistra AD, Silistra
  - Multiprofile Hospital For Active Treatment - Dr. Bratan Shukerov AD, Smolyan
  - Medical Center Hera Eood, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N. I. Pirogov EAD, Sofia
  - Diagnostic- Consultative Center Convex EOOD, Sofia
  - AES DRS Medical Center Synexus Sofia EOOD, Sofia
  - Medical Center New rehabilitation center EOOD, Stara Zagora
  - Medical Center Researchexpert OOD, Varna
  - Medical Center Tara OOD, Veliko Tarnovo
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases-Vratsa, Vratsa
- Canada (12):
  - Edmonton Respiratory Consultants, Edmonton, Alberta
  - Synergy Respiratory & Cardiac Care - Synergy Wellness Centre Location, Sherwood Park, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Dynamic Drug Advancement Ltd., Ajax, Ontario
  - Burlington Lung Clinic, Burlington, Ontario
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Inspiration Research, Toronto, Ontario
  - Dr. Syed Anees Medicine Profession Corporation, Windsor, Ontario
  - Dr Anil Dhar Professional Medicine Corporation, Windsor, Ontario
  - Clinique de pneumologie et du sommeil de Lanaudiere, Saint-Charles-Borromée, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier de l'Universite Laval, Québec
- Chile (10):
  - Centro de Estudios Clinicos, Ñuñoa
  - Centro Respiratorio Integral LTDA. (CENRESIN), Pavie Gallegos
  - Centro de Investigaciones Medicas Respiratorias CIMER, Providencia
  - Sociedad Médica SyG SpA, Providencia
  - Enroll SpA - PPDS, Providencia
  - Centro Internacional de Estudios Clínicos (CIEC), Santiago
  - Centro de Investigacion del Maule, Talca
  - Hospital Carlos Van Buren, Valparaíso
  - Centro de Investigacion de Enfermedades Respiratorias e Inmunologicas, Viña del Mar
  - Fundacion Medica San Cristobal, Vitacura
- China (36):
  - Anhui Chest Hospital, Hefei, Anhui
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - The First Hospital of Changsha, Changsha, Hunan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Huadong Hospital Affiliated of Fudan University, Shanghai, Shanghai Municipality
  - Beijing Hospital, Beijing
  - Beijing Chaoyang Hospital Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Beijing Jingmei Group General Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Third Hospital of Changsha, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Chengdu Fifth People's Hospital, Chengdu
  - The Southwest Hospital of Army Medical University, Chongqing
  - Army Medical Center of PLA(Daping Hospital), Chongqing
  - Affiliated Hospital of Guangdong Medical University, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - Huizhou Central People's Hospital, Huizhou
  - The First People's Hospital of Lian Yun Gang, Lianyungang
  - Taizhou Hospital of Zhejiang Province, Linhai
  - Jiangxi Provincial People's Hospital, Nanchang
  - Zhongda Hospital Affiliated to Southeast University, Nanjing
  - Tianjin Medical University General Hospital, Tianjin
  - Wuxi People's Hospital, Wuxi
  - Jiangyin People's Hospital, Wuxi
  - Xi'an International Medical Center Hospital, Xi'an
  - Zhongshan Hospital Xiamen University, Xiamen
  - Xinxiang First People's Hospital, Xinxiang
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai
  - Zigong First People's Hospital, Zigong
- Czechia (10):
  - Plicní ambulance MUDr. I. Cierná Peterová s.r.o., Brandýs nad Labem-Stará Boleslav
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - MediTrial s.r.o., Jind?ich?v Hradec
  - Plicni Ambulance Kralupy nad Vltavou, Kralupy nad Vltavou
  - Odborna plicni ambulance Opava s.r.o, Opava
  - Ordinace chorob plicních s.r.o., Prague
  - AES - DRS - Synexus Czech s.r.o., Prague
  - KASMED s.r.o., Tábor
  - Nemocnice Tabor, a.s., Tábor
  - Plicni stredisko Teplice s.r.o., Teplice
- Denmark (6):
  - Aalborg Universitetshospital, Aalborg
  - Gentofte Hospital, Hellerup
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense C
  - Sjaellands Universitetshospital, Roskilde, Roskilde
  - Sygehus Lillebælt, Vejle, Vejle
- France (6):
  - Clinique de l'Europe, Amiens
  - Hôpital de La Croix Rousse, Lyon
  - Hopital Saint Joseph - Marseille, Marseille
  - Hopital Pasteur II, Nice
  - Hopital Haut Leveque, Pessac
  - Nouvel Hopital Civil - CHU Strasbourg, Strasbourg
- Germany (29):
  - Zentrum fuer Pneumologie, Onkologie und Schlafmedizin am Diako, Augsburg
  - Gemeinschaftspraxis fuer Herz und Lunge am Bruderw, Bamberg
  - KPPK Studienzentrum Kroker-Schmidt, Bendorf
  - Studienpraxis Berlin-Brandenburg, Berlin, Berlin
  - Praxis fur Kardiologie und Pneumologie Dr. med. Karin Forster, Berlin
  - MECS Research GmbH, Berlin
  - AES - DRS - Synexus Berlin Research Centre, Berlin
  - Clinical Studies Pankow, Berlin
  - Lungenzentrum Darmstadt, Darmstadt
  - MVZ Jung GbR - Deggingen, Deggingen
  - Medizentrum Essen Borbeck, Essen
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Praxis Dr med Claus Keller, Frankfurt am Main
  - ME Clinical Respiratory Research Hamburg GmbH, Hamburg
  - Pneumologicum, Hanover
  - University Clinic Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Asklepios MVZ Bayern GmbH, Landsberg
  - Salvus-Klinische Studien GmbH, Leipzig
  - BAG Prof. Dr. G. Hoheisel Dr. A. Bonitz, Leipzig
  - KLB Gesundheitsforschung Lubeck GmbH, Lübeck
  - SMO.MD GmbH, Magdeburg
  - IKF Pneumologie Mainz, Mainz
  - Praxis für Pneumologie Dr. Silke Mronga & Dr. Lukas Jerrentrup, Marburg
  - Praxis Dr. med. Jan Feimer, München
  - Institut fur klinische Forschung GmbH, Neu-Isenburg
  - Studienzentrum Dr Med Schlenska, Peine
  - framol-med GmbH, Rheine
  - RoMed Klinikum Rosenheim-Pettenkoferstr. 10, Rosenheim
- Greece (6):
  - Evangelismos General Hospital of Athens, Athens
  - Navy Hospital of Athens, Athens
  - Iatriko Palaiou Falirou, Athens
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Tuen Mun Hospital, Hong Kong, Hong Kong
- Obudai Egeszsegugyi Centrum Kft.-Budapest, Budapest, Hungary
- India (12):
  - Paarthiv Lung Care Center, Hyderabad, Andhra Pradesh
  - Yashoda Hospitals Hitec City, Hyderabad, Andhra Pradesh
  - ESIC Medical College and Hospital - Faridabad, Faridabad, Haryana
  - Karnataka Institute of Medical Sciences (KIMS), Hubbali, Hubli, Karnataka
  - Shree Hospital And Critical Care Centre, Nagpur, Maharashtra
  - Kothrud Hospital, Pune, Maharashtra
  - Jawaharlal Nehru Medical College (JNMC), Ajmer, Rajasthan
  - Sawai Man Singh Hospital and Medical College, Jaipur, Rajasthan
  - Maharaja Agrasen Super Speciality Hospital, Jaipur, Rajasthan
  - Jawaharlal Nehru Medical College (JNMC), Aligarh, Uttar Pradesh
  - Apollo Spectra Hospital, Kanpur, Uttar Pradesh
  - MV Hospital and Research Centre, Lucknow, Uttar Pradesh
- Israel (13):
  - Assuta Ashdod Medical Center, Ashdod
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Centre, Beersheba
  - Shamir Medical Center Assaf Harofeh, Be’er Ya‘aqov
  - Rambam Medical Center - PPDS, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petach Tiqwa
  - Sheba Medical Center - PPDS, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Italy (5):
  - Azienda Ospedaliera Dei Colli, Napoli, Campania
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant' Anna, Cona, Ferrara, Emilia-Romagna
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Lombardy
  - Azienda Ospedaliero Universitaria Policlinico G.Rodolico - San Marco, Catania, Sicily
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Sicily
- Japan (26):
  - Japan Community Health Care Organization Hokkaido Hospital, Toyohira-ku, Sapporo City, Hokkaido
  - Matsusaka City Hospital, Matsusaka-Shi, Mie-ken
  - Shizuoka City Shizuoka Hospital, Shizuoka-Shi Aoi-Ku, Shizuoka
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Fukuwa Clinic, Chūō
  - Nishi Fukuoka Hospital, Fukuoka-Shi Nishi-Ku
  - Fukushima Medical University Hospital, Fukushima
  - National Hospital Organization Kyoto Medical Center, Fushimi-ku, Kyoto
  - Terada Respiratory and Internal Clinic, Himeji
  - Hiroshima Prefectural Hospital, Hiroshima
  - National Hospital Organization Minami Kyoto Hospital, Jōyō
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa
  - Sagamihara National Hospital, Kanagawa
  - Osaka-Minami Medical Center, Kawachinagano-Shi
  - Kishiwada City Hospital, Kishiwada-Shi
  - Juntendo Tokyo Koto Geriatric Medical Center, Kōtō City
  - National Hospital Organization Okayama Medical Center, Okayama
  - Okayama Rosai Hospital, Okayama-Shi Minami-ku
  - Omuta National Hospital, Omuta
  - Idaimae Minami 4-Jo Internal Medicine, Sapporo-shi Chuo-ku
  - Japanese Red Cross Medical Center, Shibuya-ku
  - Kamei Internal Medicine and Respiratory Clinic, Takamatsu
  - Nagata Hospital, Yanagawa
  - Yokohama City University Medical Center, Yokohama
  - Showa University Fujigaoka Hospital, Yokohama-shi Aoba-ku
  - National Hospital Organization - Yokohama Medical Center, Yokohama-Shi Totsuka-Ku
- Kenya (5):
  - KEMRI-MTWAPA Clinical Trial Site, Kilifi
  - Clinical Research Health Network (CREA-N), Machakos
  - KEMRI CRDR Clinical Research Clinic Nairobi, Nairobi
  - University of Nairobi Clinical Research Centre, Nairobi
  - Center for Research In Tropical Medicine and community development, Thika
- Latvia (4):
  - Daugavpils Regional Hospital, Daugavpils
  - Pauls Stradins Clinical University Hospital, R?ga
  - Riga 1st Hospital, Riga
  - ConsiliumMedicum, Riga
- Mexico (4):
  - CICUM San Miguel, Americana, Jalisco
  - Instituto Jalisciense de Investigacion Clinica S.A. de C.V., Santa Cecilia, Jalisco
  - Unidad Medica de Occidente, Guadalajara
  - Unidad de Investigacion Clinica En Medicina (Udicem) S.C., Monterrey
- Netherlands (5):
  - Meander Medisch Centrum, Amersfoort
  - Amphia Ziekenhuis, Breda
  - Catharina Hospital, Eindhoven
  - Dijklander Ziekenhuis - loc Hoorn, Hoorn
  - Isala Klinieken, Zwolle
- New Zealand (7):
  - P3 Research - Kapiti - PPDS, Waikanae, Wellington Region
  - Greenlane Clinical Centre, Auckland
  - NZ Respiratory & Sleep Institute, Auckland
  - Aotearoa Clinical Trials Trust, Auckland
  - Canterbury Respiratory Research Group, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
- Peru (4):
  - Clinica Providencia (Inverconsult Sociedad Anonima) - PPDS, San Miguel, Lima region
  - Clinica Internacional - PPDS, Lima
  - Medicentro Biociencias Peru S.R.L., Lima
  - Clinica Ricardo Palma - PPDS, San Isidro
- Philippines (7):
  - Manila Central University-Filemon D Tanchoco Medical Foundation, Caloocan
  - CARE CT Group Inc., Dasmariñas
  - Healthlink Medicalsurgicaldental Clinic and Diagnostic Center, Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - Mary Mediatrix Medical Center, Lipa City
  - Philippine Heart Center, Quezon City
  - Quirino Memorial Medical Center, Quezon City
- Poland (36):
  - Lekarze Specjalisci J. Malolepszy i Partnerzy, Wroclaw, Lower Silesian Voivodeship
  - AppleTreeClinics Network Sp. z o.o., Lodz, Lódzkie
  - Prywatny Gabinet Lekarski Ginekologia i Poloznictwo Ultrasonografia Prof. Jacek Suzin, Lodz, Lódzkie
  - Centrum Medycyny Oddechowej Mroz sp. j., Bia?ystok
  - Vitamed Galaj i Cichomski sp.j., Bydgoszcz
  - Medical Center Kermed, Bydgoszcz
  - Centrum Medyczne Bydgoszcz- PRATIA - PPDS, Bydgoszcz
  - Centrum Medyczne Lukamed Joanna Luka-Wendrowska, Chojnice
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Centrum Medyczne CLW-med Aneta Cichomska , Joanna Luka -Wendrowska, Grudzadz
  - Centrum Medyczne Katowice - PRATIA - PPDS, Katowice
  - Indywidualna Specjalistyczna Praktyka Lekarska lek., Kielce
  - Centrum Medyczne ALL-MED, Krakow
  - Diamond Clinic, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Medyczne ProMiMed sp z o.o. sp.k., Krakow
  - Praktyka Lekarska Adam Smialowski, Ksawerów
  - AES - DRS - Synexus Polska Sp. Z o.o. Oddzial w Lodzi, Lodz
  - ETG Lodz, Lodz
  - Clinical Best Solutions - Lublin, Lublin
  - NZOZ Przychodnia Alergologiczno-pulmonologiczna, Lublin
  - ETG Lublin, Lublin
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól
  - Ostrowieckie Centrum Medyczne Spolka Cywilna Anna Olec-Cudzik, Ostrowiec Swietokrzysk
  - Centrum Alergologii Teresa Hofman, Poznan
  - ABC-Pulmo NZOZ Agnieszka Dobielska, Jaroslaw Dobie, Radom
  - EMED Centrum Uslug Medycznych Ewa Smialek, Rzeszów
  - ETG Siedlce, Siedlce
  - Centrum Medyczne KARDIOTEL, Sopot
  - Kiepury Clinic, Sosnowiec
  - PULMAG Grzegorz Gasior Marzena Kociolek Spolka Cywilna, Sosnowiec
  - Gabinet Pulmonologii i Diagnostyki Chorob Alergicznych Dorota Malosek, Szczecin
  - CenterMed Bandrowskiego, Tarnów
  - Viltis Medica Specjalistyczna Praktyka Lekarska Lek. Med. Agata Kot, Trzebnica
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroc?aw
  - Dobrostan Gabinety Lekarskie, Wroc?aw
- Allianze Pulmonary Research LLC, Guaynabo, Puerto Rico
- Romania (4):
  - Neomed Out-Patient Treatment and Diagnosis Medical Center SRL, Brasov
  - Dr. Victor Babes Foundation, Bucharest
  - Leon Daniello Pneumophthisiology Clinical Hospital, Cluj-Napoca
  - Sf. Ioan cel Nou Emergency County Hospital, Suceava
- South Africa (15):
  - Johese Clinical Research, City of Tshwane, Gauteng
  - Iatros International, Bloemfontein
  - University of Cape Town Lung Institute, Cape Town
  - Dr. Ismail Abdullah Private Practice, City of Cape Town
  - Newtown Clinical Research Centre, City of Johannesburg
  - Clinical Trial Systems, City of Tshwane
  - St Augustines Hospital, Durban
  - Lakeview Hospital, Ekurhuleni
  - Dr A.C Wilhase practice-Reimed, Ekurhuleni
  - CLINRESCO, ARWYP Medical Suites, Ekurhuleni
  - Langeberg Clinical Trials, Kraaifontein
  - Medicross Pretoria West, Jongaie Research, Pretoria
  - AES - DRS - Synexus Watermeyer Clinical Research Centre, Pretoria
  - AES - DRS - Synexus - Helderberg Clinical Research Centre, Somerset West
  - Dr Yacoob AK Private Practice, Welkom
- South Korea (13):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Yeungnam University Hospital, Daegu
  - CHA Bundang Medical Center, Gyeonggi-do
  - Catholic Univ. of Incheon St.Mary's Hospital, Incheon
  - Chonbuk National University Hospital, Jeollabuk-do
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (15):
  - Hospital de Merida, Mérida, Badajoz
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, LA Coruna
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Vithas Xanit International Hospital, Benalmádena Costa, Malaga
  - Hospital de La Ribera, Alzira, Valencia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (5):
  - Fysikalisk Medicin i Stockholm AB, Lidingö
  - Clinical Trial Consultants - Linkoping, Linköping
  - PharmaSite, Malmo
  - ProbarE i Stockholm AB, Stockholm
  - Akardo AB, Stockholm
- Zurcher Reha Zentren Wald, Zurich, Switzerland
- Taiwan (6):
  - Changhua Christian Hospital, Chang-hua
  - Kaohsiung Medical University Hospital, Kaoshiung City
  - Far East Memorial Hospital, New Taipei City
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Thailand (2):
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Central Chest Institute of Thailand, Muang
- Turkey (Türkiye) (3):
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Kirikkale Universitesi Tip Fakultesi Hastanesi, Kırıkkale
  - Rize Recep Tayyip Erdogan University Training and Research Hospital, Rize Merkez
- United Kingdom (14):
  - Guys Hospital, London, Middlesex
  - AES - DRS - Synexus Scotland Clinical Research Centre, Bellshill
  - Bradford Royal Infirmary, Bradford
  - Addenbrookes Hospital, Cambridge
  - AES - DRS - Synexus Wales Clinical Research Centre, Cardiff
  - Royal Primary Care - Ashgate Manor, Chesterfield
  - AES - DRS - NW Consortium Lancashire, Chorley
  - Castle Hill Hospital, Cottingham
  - AES - DRS - Synexus Midlands Clinical Research Centre, Edgbaston
  - AES - DRS - Synexus Hexham Clinical Research Centre, Hexham
  - Glenfield Hospital, Leicester
  - AES - DRS - NW Consortium Merseyside, Liverpool
  - Velocity Clinical Research North London - Percy Road - PPDS, London
  - Queen Anne Street Medical Centre, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing